CLINICAL TRIAL: NCT02896530
Title: Arterial Thrombosis and Inflammatory Bowel Disease: a Series of 6 Cases and Literature Review
Acronym: TAMICI
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: TAMICI
Record Dates: First submitted 2016-08-31; First posted 2016-09-12 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Arterial Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention. Description study

SUMMARY:
Vascular complications in patients with inflammatory bowel disease (IBD), comprising mainly Crohn's disease (CD) and ulcerative colitis (UC), representing 2% extra-intestinal complications. In over 60% of cases, these vascular complications of deep venous thrombosis (DVT) or pulmonary embolism (PE). Several studies have shown that patients with IBD have a risk of venous thromboembolic disease (VTE) increased from 1.5 to 3.5. This risk is closely related to disease activity.

DETAILED DESCRIPTION:
Vascular complications in patients with inflammatory bowel disease (IBD), comprising mainly Crohn's disease (CD) and ulcerative colitis (UC), representing 2% extra-intestinal complications. In over 60% of cases, these vascular complications of deep venous thrombosis (DVT) or pulmonary embolism (PE). Several studies have shown that patients with IBD have a risk of venous thromboembolic disease (VTE) increased from 1.5 to 3.5. This risk is closely related to disease activity.

However, the association between IBD and arterial thromboembolic events such as cases of myocardial infarction, stroke, aortic thrombus, mesenteric ischemia, peripheral arterial disease and members senior, was described less and remains a subject of debate. These arterial complications occur in young subjects accountability of IBD remains debated, and no clear pathophysiology. Here the investigators describe a series of 6 cases of patients with IBD who developed severe arterial complications, and whose cause was retained digestive inflammatory underlying disease.

This study is report of six (6) cases that will be described

ELIGIBILITY:
Inclusion Criteria:

* Patients with arterial Thrombosis and Inflammatory Bowel Disease admitted in Paris Saint Joseph Hospital

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with arterial Thrombosis and Inflammatory Bowel Disease
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2015-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Assessment of change of the number of thromboembolic events or venous or arterial | Month 6, year 2

SECONDARY OUTCOMES:
Assessment of the relevance of anti thrombosis treatment | Month 6, year 2
  Is the anti thrombosis treatment adequate or have been changed during the monitoring? The answer to this question should be :yes or no

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided